CLINICAL TRIAL: NCT02256332
Title: Effect of Plant-based Ingredient on Post Prandial Glucose in Untreated Type II Diabetes Patients
Brief Title: Plant-based Ingredient on Post Prandial Glucose in Type II Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FDS-NAA-1633
Record Dates: First submitted 2014-09-30; First posted 2014-10-03 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose plant based ingredient (Active Comparator): Reference food with low dose of plant based ingredient
  Interventions: Dietary Supplement: Low dose plant based ingredient
- High dose plant based ingredient (Active Comparator): Reference food with high dose of plant based ingredient
  Interventions: Dietary Supplement: High dose plant based ingredient
- Reference food format (Placebo Comparator): Reference food without plant-based ingredient
  Interventions: Dietary Supplement: Reference food format

INTERVENTIONS:
Dietary Supplement: Low dose plant based ingredient — Reference food with low dose of plant based ingredient
  Arms: Low dose plant based ingredient
Dietary Supplement: High dose plant based ingredient — Reference food with high dose of plant based ingredient
  Arms: High dose plant based ingredient
Dietary Supplement: Reference food format — Reference food without plant-based ingredient
  Arms: Reference food format

SUMMARY:
Effects of a plant based ingredient on blood glucose in Type II diabetes patients.

DETAILED DESCRIPTION:
The study is designed to determine the extend to which a plant based ingredient in a food format affects blood glucose responses in untreated Type II diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers with confirmed Type II diabetes not treated with pharmaceutical-based glucose lowering treatment for past three months (controlled solely through diet and exercise);
* Age ≥ 20 and ≤ 65 year at screening;
* Body Mass Index (BMI) between ≥18 and ≤ 32 kg/m2;
* HbA1c ≥48 mmol/mol and ≤53 mmol/mol (≥ 6.5% and ≤ 7.0%). At discretion of the study physician, subjects with HbA1c >53 mmol/mol and <58 mmol/mol (>7.0% and < 7.5%) controlled solely through diet and exercise are also allowed to participate.

Exclusion Criteria:

* Being an employee of Unilever or research site;
* Chronic smokers, tobacco chewers and drinkers;
* No medication, including vitamins and tonics, except for cholesterol, as determined by the physician;
* Reported weight loss/gain ≥ 10% of body weight in the 6 months preceding screening;
* Allergy to any food or cosmetics;
* If female, not being pregnant or planning pregnancy during the study period;
* If female, lactating or has been lactating for 6 weeks before pre-study investigation and/or during the study period.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Post prandial blood glucose positive incremental area under the curve | 120 minutes

SECONDARY OUTCOMES:
Post prandial insulin area under the curve | 120 minutes

OTHER OUTCOMES:
Post prandial blood glucose positive incremental area under the curve | 180 and 240 minutes
Post prandial insulin area under the curve | 180 and 240 minutes
Glucose levels in urine | 240 minutes
Intestinal discomfort | 240 minutes
  Intestinal discomfort will be evaluated by a paper and pen questionnaire in the subject's native language directed to intestinal symptoms (nausea, flatulence, bloating and abdominal pain).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ketul Modi, MBBS, Principal Investigator — Lambda Therapeutics Research Ltd (LTRL); Dr Shrikant V Deshpande, Principal Investigator — Ashirwad Hospital and Research Centre, THANE , MAHARASHTRA
Locations (2):
- India (2):
  - Ashirwad Hospital and Research Centre, THANE , MAHARASHTRA, Thane, Maharashtra
  - Lambda Therapeutics Research Ttd (LTRL), Ahemdabad